CLINICAL TRIAL: NCT00452738
Title: The Effect of Pre Surgery Dog Visits on Post Surgery Consumption of Pain Medication
Acronym: Dog
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left university. Did not start study
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006036
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2008-01

CONDITIONS: Post Tonsillectomy Pain
Keywords: animal-assisted intervention; pre surgery anxiety; post surgery pain medication consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Therapy dog
Behavioral: Costumed character
Behavioral: Parents-only

SUMMARY:
The objective of this study is to examine the effects of pre surgery dog visits as compared to a costumed character or parents-only on the consumption of pain medication after surgery. It is hypothesized that pre surgery dog visits will reduce post surgical stress and anxiety.

DETAILED DESCRIPTION:
Recent research has revealed that children who are highly anxious prior to surgery experienced more problems post surgery. These problems included reporting of more pain and requested more pain medication during hospitalization and home follow up. Consumption of pain medication may not be the optimal pain management program. In contrast, numerous human-animal interaction studies have shown that animals tend to have a calming effect on people, reduce stress, and lesson anxiety. Therefore, the primary objective of this study is to examine the effect of pre surgery dog visits as compared to a costumed character or parents-only on the consumption of pain medication after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy and Adenoidectomy (T/A)
* 4-7 years old
* Prescribed codeine and/or analgesics for postoperative pain

Exclusion Criteria:

* Participant must not be afraid of dogs, or allergic to animal dander
* Chronic medical conditions other than T/A
* Developmentally delayed
* On psychotropic medications

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-04; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Bieri Faces Scale upon arrival, after intervention, and at discharge
Modified Yale Preoperative Anxiety Scale upon arrival, after intervention, and in surgical preparation room

CONTACTS AND LOCATIONS:
Overall Officials: Sherril M Stone, PhD, Principal Investigator — Oklahoma State University Center for Health Sciences; Stan Sherman, DO, Principal Investigator — Oklahoma State University Center for Health Sciences; Chaunda Capers, BS, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State University Surgi-Center, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Bieri D, Reeve RA, Champion DG, Addicoat L, Ziegler JB. The Faces Pain Scale for the self-assessment of the severity of pain experienced by children: development, initial validation, and preliminary investigation for ratio scale properties. Pain. 1990 May;41(2):139-150. doi: 10.1016/0304-3959(90)90018-9. PMID 2367140
- [Background] Brodie SJ, Biley FC, Shewring M. An exploration of the potential risks associated with using pet therapy in healthcare settings. J Clin Nurs. 2002 Jul;11(4):444-56. doi: 10.1046/j.1365-2702.2002.00628.x. PMID 12100640
- [Background] Caprilli S, Messeri A. Animal-Assisted Activity at A. Meyer Children's Hospital: A Pilot Study. Evid Based Complement Alternat Med. 2006 Sep;3(3):379-83. doi: 10.1093/ecam/nel029. Epub 2006 Apr 2. PMID 16951723
- [Background] Center for Disease Control (CDC) (2006). Hand Sanitizer Alert. www.cdc.gov/ncidod/eid/vol12no03/05-0955.htm.
- [Background] Delta Society (2006). About Animal-assisted activities & Animal-assisted therapy. www.deltasociety.org/AnimalsAAAAbout.htm.
- [Background] Denver Children's Hospital. (1990). Facts: Prescription pet program. Denver, CO: Author.
- [Background] Feld LH, Negus JB, White PF. Oral midazolam preanesthetic medication in pediatric outpatients. Anesthesiology. 1990 Nov;73(5):831-4. doi: 10.1097/00000542-199011000-00006. PMID 2240672
- [Background] Fry WF Jr. The physiologic effects of humor, mirth, and laughter. JAMA. 1992 Apr 1;267(13):1857-8. doi: 10.1001/jama.267.13.1857. No abstract available. PMID 1545471
- [Background] Golden L, Pagala M, Sukhavasi S, Nagpal D, Ahmad A, Mahanta A. Giving toys to children reduces their anxiety about receiving premedication for surgery. Anesth Analg. 2006 Apr;102(4):1070-2. doi: 10.1213/01.ane.0000198332.51475.50. PMID 16551900
- [Background] Green Chimneys (2006). www.greenchimneys.com/about.htm.
- [Background] Johnson RA, Odendaal JS, Meadows RL. Animal-assisted interventions research: issues and answers. West J Nurs Res. 2002 Jun;24(4):422-40. doi: 10.1177/01945902024004009. PMID 12035914
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Mayes LC, Caramico LA, Silver D, Spieker M, Nygren MM, Anderson G, Rimar S. Parental presence during induction of anesthesia. A randomized controlled trial. Anesthesiology. 1996 May;84(5):1060-7. doi: 10.1097/00000542-199605000-00007. PMID 8623999
- [Background] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Gaal D, Wang SM, Mayes LC. Interactive music therapy as a treatment for preoperative anxiety in children: a randomized controlled trial. Anesth Analg. 2004 May;98(5):1260-6, table of contents. doi: 10.1213/01.ane.0000111205.82346.c1. PMID 15105197
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Moody WJ, King R, O'Rourke S. Attitudes of paediatric medical ward staff to a dog visitation programme. J Clin Nurs. 2002 Jul;11(4):537-44. doi: 10.1046/j.1365-2702.2002.00618.x. PMID 12100650
- [Background] Odendaal JS. Animal-assisted therapy - magic or medicine? J Psychosom Res. 2000 Oct;49(4):275-80. doi: 10.1016/s0022-3999(00)00183-5. PMID 11119784
- [Background] Peterson L, Ridley-Johnson R. Pediatric hospital response to survey on prehospital preparation for children. J Pediatr Psychol. 1980 Mar;5(1):1-7. doi: 10.1093/jpepsy/5.1.1. No abstract available. PMID 7452418
- [Background] Piaget, J. (1952). The origins of intelligence in children. International Universities Press. New York: NY.
- [Background] Roosevelt M. Canine candy stripers. Time. 2001 Aug 6;158(5):52-3. No abstract available. PMID 11499222
- [Background] Saint Mary's Hospital. (1995). Pet therapy on PEDS unit: Happiness is a warm puppy. Rochester: MN.
- [Background] Santrock, John W. (2001). Child development. Ninth Edition, 2, 36-37.
- [Background] Serpell, J. A. (2000). Creatures of the unconscious: Companion animals as mediators. In A. L. Podberscek, E. S. Paul & J. A. Serpall (Eds.), Companion animals and us: Exploring the relationship between people and pets (pp. 108-124). New York: Cambridge University Press.
- [Background] Sobo EJ, Eng B, Kassity-Krich N. Canine visitation (pet) therapy: pilot data on decreases in child pain perception. J Holist Nurs. 2006 Mar;24(1):51-7. doi: 10.1177/0898010105280112. PMID 16449747
- [Background] Spielberger C. D. (1983). Manual for the State-Trait Anxiety Inventory (STAI: Form Y), Consulting Psychologists Press, Palo Alto: CA.
- [Background] Vagnoli L, Caprilli S, Robiglio A, Messeri A. Clown doctors as a treatment for preoperative anxiety in children: a randomized, prospective study. Pediatrics. 2005 Oct;116(4):e563-7. doi: 10.1542/peds.2005-0466. PMID 16199685
- [Background] Viitanen H, Annila P, Viitanen M, Tarkkila P. Premedication with midazolam delays recovery after ambulatory sevoflurane anesthesia in children. Anesth Analg. 1999 Jul;89(1):75-9. doi: 10.1097/00000539-199907000-00014. PMID 10389782
- [Background] Weisenberg M, Raz T, Hener T. The influence of film-induced mood on pain perception. Pain. 1998 Jun;76(3):365-375. doi: 10.1016/S0304-3959(98)00069-4. PMID 9718255
- [Result] Arkow, P. (1993). Pet therapy: A study and resource guide for the use of companion animals in selected therapies (7th ed.). Humane Society of the Pikes Peak Region. Colorado Springs: CO
- [Result] Barba, B. (1995). A critical review of research on the human/companion animal relationship 1988-1993. Anthrozoos, 8(1), 9-15.
- [Result] Bell, J. R. (2006). Visitation dogs carry C. difficile, MRSA, Salmonella. Family Practice News, 28.
- [Result] Donowitz LG. Pet therapy. Pediatr Infect Dis J. 2002 Jan;21(1):64-6. doi: 10.1097/00006454-200201000-00016. No abstract available. PMID 11791104
- [Result] Friedman, E., Thomas, S. A., & Eddy, T. J. (2000). Companion animals and human health: Physical and cardiovascular influences. In A. L. Podberscek, E. S. Paul, & J. A. Serpell (Eds), Companion animals and use: Exploring the relationship between people and pets (pp. 125-142). New York: Cambridge University Press.
- [Result] Jalongo, M. R. (2004). The world's children and their companion animals: Developmental and educational significance of the child/pet bond. Association for Childhood Education International. Olney: ND.
- [Result] Jalongo, M. R., Astorino, T., & Bomboy, N. (2004). Canine Visitors: The Influence of therapy Dogs on Young Children's Learning and Well-Being in Classrooms and Hospitals. Early Childhood Education Journal, 32(1), 9-16.
- [Result] Kaminski, M., Pellino, T., & Wish, J. (2002). Play and Pets: The Physical and Emotional Impact of Child-Life and Pet Therapy on Hospitalized Children. Children's Health Care, 31(4), 321-335.
- [Result] Mallon, G. (1994). Some of our best therapists are dogs. Child and Youth Care Forum, 23, 89-101.
- [Result] Melson, G. F. (2001). Why The Wild Things Are. Harvard University Press. Cambridge: MA.
- [Result] Pembrook, L. (2005). Distraction with handheld video game is an effective anxiolytic, Anesthesiology News, 31(3), 4-6.
- [Result] Schantz, (1990). Reviews and research reports; Preventing potential health hazards incidental to the use of pets in therapy. Anthrozoos, 4(1), 114-123.